CLINICAL TRIAL: NCT07159204
Title: The Paclitaxel Polymer Micellar Based Combined Immunotherapy for the Posterior Line Treatment of Advanced Bile Tract Cancer
Brief Title: Paclitaxel mIcelle Later-line cOmbined immunoTherapy for Biliary Tract Cancer
Acronym: PILOT-BTC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K6146
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel polymer micelle immunocombination (Experimental)
  Interventions: Drug: Paclitaxel polymer micelle immunocombination

INTERVENTIONS:
Drug: Paclitaxel polymer micelle immunocombination — Paclitaxel polymer micelle immunocombination

SUMMARY:
After the standard first-line treatment, the treatment regimen was adjusted to a paclitaxel polymer micellar-based immunotherapy combination regimen

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and agreed to sign the written informed consent, with good compliance and follow-up, and were at least 18 years old at the time of signing the informed consent, regardless of gender.
* Patients with advanced biliary carcinoma diagnosed by imaging and histology as unresectable, recurrent, locally advanced, or with metastatic lesions are defined as stage IIIA or above according to the AJCC-8 staging system, including intrahepatic or extrahepatic cholangiocarcinoma and gallbladder cancer. No more than 2 organs metastasized, including liver, lung, bone, and brain.
* Radical surgery/local treatment, including focal excision, ablation, transcatheter arterial chemoembolization, hepatic arterial infusion chemotherapy, and radiotherapy, is not appropriate for at least 4 weeks prior to baseline assessment, or for disease progression thereafter. All acute toxic effects during local treatment must be ≤CTCAE5.0 grade 1.
* Patients were intolerant or failed for ≥1 month after first-line systemic therapy, required palliative care, and patient adverse events were controlled (NCI-CTCAE≤ Grade I).
* At least one measurable lesion (a spiral CT scan of a measurable lesion ≥10mm or an enlarged lymph node ≥15mm, as required by RECIst version 1.1).
* The ECOG score in the first week of enrollment was 0-1. Survival was expected to be ≥3 months as assessed by the investigators.
* Active hepatitis B and C patients are required to receive relevant antiviral therapy, HBV-DNA < 2000 IU/ml (< 104 copies /ml), and have received anti-HBV therapy for at least 14 days prior to study entry and continue treatment during treatment. HCV RNA-positive patients must receive antiviral therapy according to standard local treatment guidelines and have liver function within CTCAE grade 1 elevation.
* Hematology and organ function are adequate, based on the following laboratory results obtained within 14 days prior to initiation of investigational therapy (unless otherwise indicated)
* Any clinically significant biliary obstruction should be resolved before randomization.
* Adequate renal function: creatinine ≤1.5×ULN, or creatinine clearance >50mL/min
* Women who are fertile: agree to abstain from sex (abstain from heterosexual intercourse) or use a contraceptive method with an annual contraceptive failure rate of < 1% during treatment and for at least 6 months after the last dose.
* Men: agree to abstain from sex (no heterosexual intercourse) or use contraception, and agree not to donate sperm.

Exclusion Criteria:

* Those who have previously received treatment with immune checkpoint inhibitors, lenvatinib or paclitaxel, or are known to be allergic to or intolerant to immune checkpoint inhibitors, lenvatinib or paclitaxel and their components
* Any systemic anti-tumor treatment received within the three months prior to participating in the study, including but not limited to intravenous infusion and/or oral chemotherapy, targeted drugs, antibody drugs and traditional Chinese medicines with known anti-cancer effects.
* The patient is undergoing approved or under-development systemic anti-cancer therapies, including chemotherapy, biological immunotherapy, targeted therapy, or traditional Chinese medicine therapy with clear indications. Treatment is allowed 4 weeks before randomization.
* The histopathological results show a mixture of liver cancer, squamous cell carcinoma or sarcoma cell components, or ampullary carcinoma.
* Accompanied by other malignant tumors, but having had other uncured malignant tumors in the past (within 5 years) or simultaneously.
* Significant digestive tract diseases: Pre-existing or existing grade 3 or above digestive tract fistula or non-digestive tract fistula as per CTCAE 5.0 criteria. There is evidence or history of bleeding mechanism disorders such as a history of gastrointestinal bleeding within the last 6 months, or a clear tendency of gastrointestinal bleeding, or a gastrointestinal bleeding event of grade ≥3 (CTCAE 5.0).
* Cardiovascular and cerebrovascular diseases with significant clinical significance Including but not limited to having experienced acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accident or transient ischemic attack within 6 months prior to enrollment, congestive heart failure, arrhythmia requiring treatment, hypertension that has not been well controlled after antihypertensive drug treatment, and a history of thromboembolism (including stroke and/or transient ischemic attack) within the last 6 months.
* Liver and kidney insufficiency: Liver insufficiency: Characterized by jaundice, ascites and/or bilirubin >3×ULN. Renal insufficiency: Creatinine ratio >3.5g/24 hours, urine routine showing urine protein ≥++ or confirmed 24-hour urine protein quantification > 1.0g, or renal failure requiring hemodialysis or peritoneal dialysis, etc. Having received treatment with a potent CYP3A4 inhibitor within 7 days before participating in the study, or having received treatment with a potent CYP3A4 inducer within 12 days before participating in the study.
* Have active autoimmune diseases or a history of autoimmune diseases or are at risk of immune diseases: Have suffered from active, known or suspected autoimmune diseases in the past two years, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, etc. Be ready or have previously received organ or allogeneic bone marrow transplantation. Alternative therapy is not considered a form of systemic treatment for participants who may have their vital organ functions affected or who have already/may need systemic immunosuppressive therapy. This clinical trial allows patients with type 1 diabetes, hypothyroidism with only hormone replacement, skin diseases that do not require systemic treatment, or those who will not relapse without external triggers to participate.
* Neurological disorders: Known or untreated brain metastases, or patients with epilepsy requiring drug treatment. Known active central nervous system metastases and/or cancerous meningitis. Subjects with previously treated brain metastases but stable brain metastasis disease (no evidence of progression on imaging at least four weeks before the first trial treatment and any neurological symptoms have returned to baseline) can participate, without evidence of new or expanded brain metastases, and without steroid use for at least 7 days before the trial treatment. However, cancerous meningitis is not included. Regardless of clinical stability, it is excluded.
* Infectious disease: Persistent infection with grade >2 (CTCAE 5.0). A known history of active tuberculosis (Mycobacterium tuberculosis). A known history of human immunodeficiency virus (HIV) infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline (≤28 days before first dose); every 6 weeks (±7 days) through Week 24 (primary analysis time point); then every 12 weeks until disease progression or start of new anticancer therapy, through study completion (up to 24 months).
  Proportion of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v1.1, assessed by investigators using contrast-enhanced abdominal CT or MRI (PET-CT may be supportive but not response-defining). Two consecutive scans ≥4 weeks apart are required to confirm response. Measure Type / Unit: Percentage of participants (%)
Adverse Events (AEs) | From first dose (Day 1) through 30 days after the last dose for AEs; serious AEs monitored through 90 days after the last dose; through study completion (up to 24 months).
  Incidence, nature, and severity of treatment-emergent adverse events graded per NCI CTCAE v5.0; includes serious AEs and AEs leading to dose modification or discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim JY, Do YR, Song HS, Cho YY, Ryoo HM, Bae SH, Kim JG, Chae YS, Kang BW, Baek JH, Kim MK, Lee KH, Park K. Multicenter Phase II Clinical Trial of Genexol-PM(R) with Gemcitabine in Advanced Biliary Tract Cancer. Anticancer Res. 2017 Mar;37(3):1467-1473. doi: 10.21873/anticanres.11471. PMID 28314319